CLINICAL TRIAL: NCT01195623
Title: Randomized Clinical Trial of Routine Preoperative Duplex Imaging Before Varicose Vein Surgery; Long-term Follow-up
Brief Title: The Long-term Value of Preoperative Duplex Before Surgery for Varicose Veins
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Uppsala University Hospital (Other)
Collaborators: Capio Research Foundation (Other); Region Stockholm (Other Government)
Responsible Party: Principal Investigator, Lena Blomgren, MD, PhD, Uppsala University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: ETKI 96-169
Record Dates: First submitted 2010-09-03; First posted 2010-09-06 (Estimated); Results first posted 2013-02-15 (Estimated); Last update posted 2013-02-15 (Estimated); Status verified 2013-02

CONDITIONS: Varicose Veins
Keywords: varicose veins; venous insufficiency; surgery; duplex; recurrence
MeSH Terms: conditions — Varicose Veins; Venous Insufficiency; Recurrence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- varicose vein surgery with preop duplex (Active Comparator): The surgeon has planned surgery for varicose veins from a clinical examination and has then the extra information available from a preoperative duplex examination to plan surgery more in detail
  Interventions: Procedure: preoperative duplex examination; Procedure: Preoperative duplex
- varicose vein surgery no preop duplex (No Intervention): The surgeon has planned surgery for varicose veins from a clinical examination only

INTERVENTIONS:
Procedure: preoperative duplex examination
  Arms: varicose vein surgery with preop duplex
Procedure: Preoperative duplex
  Arms: varicose vein surgery with preop duplex

SUMMARY:
Duplex imaging is costly and time-consuming, but is used increasingly for preoperative evaluation of varicose veins. Its value in terms of the long-term results of surgery is not clear. 293 patients (343 limbs) with primary varicose veins were randomized to operation with or without preoperative duplex imaging. Reoperation rates, clinical and duplex findings were compared at 2 months and 2 years after surgery. Routine preoperative duplex examination led to an improvement in results. However two years is a short time, and with a longer follow-up other mechanisms for recurrence may become more important, e.g. neovascularization (new vessel formation) or progression of disease, hence the value of a detailed preoperative diagnosis may be diminished. The aim of this phase of the investigation is to study the results after 8 years, in particular what mechanisms for recurrences were most important.

ELIGIBILITY:
Inclusion Criteria:

* patients with primary varicose veins

Exclusion Criteria:

* pure cosmetic complaints
* previous venous surgery or sclerotherapy
* history of suspect or manifest deep venous thrombosis
* active or healed venous ulceration
* peripheral arterial disease
* previous significant trauma to the leg
* general illness
* alcohol or drug abuse
* unable to understand information

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 293 (Actual)
Dates: Start 1997-11; Primary Completion 2003-09 (Actual); Study Completion 2010-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Capio StGörans Gospital, Stockholm, Sweden

REFERENCES:
- [Background] Blomgren L, Johansson G, Bergqvist D. Quality of life after surgery for varicose veins and the impact of preoperative duplex: results based on a randomized trial. Ann Vasc Surg. 2006 Jan;20(1):30-4. doi: 10.1007/s10016-005-9285-z. PMID 16378147
- [Background] Blomgren L, Johansson G, Dahlberg-Akerman A, Thermaenius P, Bergqvist D. Changes in superficial and perforating vein reflux after varicose vein surgery. J Vasc Surg. 2005 Aug;42(2):315-20. doi: 10.1016/j.jvs.2005.03.043. PMID 16102633
- [Result] Blomgren L, Johansson G, Bergqvist D. Randomized clinical trial of routine preoperative duplex imaging before varicose vein surgery. Br J Surg. 2005 Jun;92(6):688-94. doi: 10.1002/bjs.4983. PMID 15810046
- [Result] Blomgren L, Johansson G, Emanuelsson L, Dahlberg-Akerman A, Thermaenius P, Bergqvist D. Late follow-up of a randomized trial of routine duplex imaging before varicose vein surgery. Br J Surg. 2011 Aug;98(8):1112-6. doi: 10.1002/bjs.7579. Epub 2011 May 27. PMID 21618499
- [Derived] Blomgren L. Residual incompetent tributaries after varicose vein surgery increased the need for reintervention after 8 years. J Vasc Surg Venous Lymphat Disord. 2020 May;8(3):378-382.e1. doi: 10.1016/j.jvsv.2019.11.012. Epub 2020 Jan 25. PMID 31992538

RESULTS

PARTICIPANT FLOW:
Groups:
- Varicose Vein Surgery With Preoperative Duplex: The surgeon has planned surgery for varicose veins from a clinical examination and has then the extra information available from a preoperative duplex examination to plan surgery more in detail
- Varicose Vein Surgery Without Preoperative Duplex: The surgeon has planned surgery for varicose veins from a clinical examination only
Period: Overall Study
Arm/Group | Varicose Vein Surgery With Preoperative Duplex | Varicose Vein Surgery Without Preoperative Duplex
Started | 148 (166 legs total operated) | 145 (177 legs total operated)
Completed | 113 (127 legs) | 108 (129 legs)
Not Completed | 35 | 37
Not completed — Lost to Follow-up | 35 | 37

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Varicose Vein Surgery With Preoperative Duplex | Varicose Vein Surgery Without Preoperative Duplex | Total
Number analyzed (Participants) | 148 | 145 | 293
Age Continuous [Mean (Standard Deviation); unit: years] | 56.3 (10.6) | 52.6 (12.9) | 54 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 108 | 109 | 217
  Male | 40 | 36 | 76
Region of Enrollment [Number; unit: participants]
  Sweden | 148 | 145 | 293

OUTCOME MEASURES:

1. Primary Outcome: Rate of Re-do Surgery
Description: number of reoperations (legs) in the two treatment arms
Time Frame: 7 years mean
Population: The number of legs has been analyzed, randomized 166 legs in the duplex group and 177 in the no-duplex group
Measure: Number; unit: legs
Arm/Group | Varicose Vein Surgery With Preoperative Duplex | Varicose Vein Surgery Without Preoperative Duplex
Number analyzed (Participants) | 124 | 134
legs | 15 | 38

2. Secondary Outcome: Recurrence Rate
Description: number of recurrences in treatment arms but also nature of recurrences
Time Frame: 7 years
Population: The number of legs with recurrence of varicose veins in the saphenofemoral junction (SFJ)or saphenopopliteal junction (SPJ)
Measure: Number; unit: legs
Units Other Than Participants: legs
Arm/Group | Varicose Vein Surgery With Preoperative Duplex | Varicose Vein Surgery Without Preoperative Duplex
Number analyzed (Participants) | 85 | 87
Number analyzed (legs) | 95 | 99
legs | 13 | 46

ADVERSE EVENTS:
Arm/Group | Varicose Vein Surgery With Preoperative Duplex | Varicose Vein Surgery Without Preoperative Duplex
Serious Adverse Events (participants affected / at risk) | 0/148 | 0/145
Other Adverse Events (participants affected / at risk) | 0/148 | 0/145

LIMITATIONS AND CAVEATS:
The rate of hand-held Doppler device use was not known and may have influenced the results, however even now many Swedish surgeons plan varicose vein surgery clinical tests only

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes